CLINICAL TRIAL: NCT03960632
Title: Clinical Performance Evaluation of Malaria Pf Plus RDT and Malaria Pf/Pv Plus RDT for the Detection of Plasmodium Infections in Patients With Symptoms Suggestive of Malaria
Brief Title: Performance Evaluation of Malaria Plus RDTs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 7874-2/1
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Abbott SD Bioline Malaria Pf Plus (05FK150) and Abbott SD Bioline Malaria Pf/Pv Plus (05FK160)) — Qualitative in vitro tests for the detection of Plasmodium antigens

SUMMARY:
Since their introduction in the late 90's, rapid diagnostic tests (RDTs) have dramatically improved our ability to control malaria, but proved insufficient to support elimination efforts because of their limited sensitivity, especially for P. vivax. In addition, the spread of P. falciparum parasites lacking hrp2 gene jeopardizes the long-term use of P. falciparum-specific HRP2-based RDTs. An existing partnership between Standard Diagnostics (SD), FIND, PATH, and Bill and Melinda Gates Foundation (BMGF) is addressing these limitations by developing two novel malaria RDTs with an analytical sensitivity ten times higher than the currently available malaria RDTs: a P. falciparum-specific test targeting both the HRP2 and PfLDH antigens (Pf Plus), and a P. falciparum/P. vivax combo test additionally targeting the PvLDH antigen (Pf/Pv Plus).

These new combo tests with improved sensitivity may become promising diagnostic tools for the detection of malaria, especially in settings where current tests prove to be insufficient due to hrp2 deletion or high burden of P. vivax malaria.

In this study, the investigators will perform a prospective evaluation of Pf Plus and Pf/Pv Plus tests in malaria-endemic countries to assess their clinical performance for detection of malaria in their intended-use settings.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at the study site with fever (axillary temperature ≥37.5°C) or a history of fever during the preceding 72 hours period
* Presence of symptoms and signs other than fever suggestive of malaria
* Aged 5 years or older
* Freely agreeing to participate by signing an informed consent form (adults aged 18 and older and parent/legal guardian of a child) and providing assent (children aged 13-17)
* Willing to provide finger prick blood sample at enrolment

Exclusion Criteria:

* Presence of symptoms and signs of severe disease and/or central nervous system infections, as defined by WHO guidelines

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms suggestive of malaria seeking clinical care in health facilities
Sampling Method: Non-Probability Sample
Enrollment: 6546 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Estimates of clinical performance characteristics of Pf Plus | Enrolment
  Estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV, and DOR) of Pf Plus using the primary reference test (qPCR) as standard of truth for the detection of malaria in patients with symptoms suggestive of malaria
Estimates of clinical performance characteristics of Pf/Pv Plus | Enrolment
  Estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV, and DOR) of Pf/Pv Plus using the primary reference test (qPCR) as standard of truth for the detection of malaria in patients with symptoms suggestive of malaria

IPD SHARING:
Plan to Share IPD: Undecided